CLINICAL TRIAL: NCT02051517
Title: Vitreous Chemistry Analysis
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1303M30101
Record Dates: First submitted 2013-12-16; First posted 2014-01-31 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Normal Volunteers
Keywords: Virectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Vitreous fluid whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitrectomy: Subjects expected to have normal vitreous, undergoing vitrectomy surgery for medically indicated reasons.

SUMMARY:
The aim of this study is to expand the understanding of the vitreous, its solute chemistry, and the normal relationship of that chemistry to the chemistry of the systemic circulation in humans.

Sample human vitreous from patients undergoing vitrectomy surgery and compare to results of metabolic chemistry panel from subject.

Allow the research team to extract .2ml sample of the .5ml - 1.0ml vitreous that is normally extracted during a routine undiluted vitreous biopsy, a standard procedure performed for various indications. Blood draw for metabolic chemistry panel (1-2 ml).

DETAILED DESCRIPTION:
The proposed method for obtaining antemortem vitreous samples is during an otherwise scheduled vitrectomy surgery that is being performed for a medically necessary indication. Virectomy surgery is a commonly performed eye surgery during which the vitreous humor is removed from the eye. Three ports are created through the sclera for access into the eye. One port is for a light to provide illumination for visualization, one port is for the vitrector, which simultaneously aspirates the vitreous and cuts its intrinsic fibers, and one port is for an infusion line which keeps the eye inflated with saline as the vitreous humor is removed. typically the aspiration is performed automatically by the vitrectomy machine. For an undiluted vitreous biopsy, which is standard procedure performed for various indications, the technique must be slightly modified. In particular, the infusion line is not turned on initially to avoid diluting the specimen with saline fluid. The vitrector aspiration line is connected to a syringe instead of the vitrectomy machine, and the syringe is used to both manually provide the aspiration and to collect the undiluted specimen. As soon as an adequate volume is collected, the infusion line is turned on and the aspiration line is reconnected to the vitrectomy machine. Volumes of 0.5 to 1.0 ml are routinely collected with this technique.

Subjects will be enrolled from adult patient already undergoing vitrectomy surgery for various retinal conditions. Only one eye per subject will be enrolled and the enrollment target for the first year is 50 subjects.

Specimens would be obtained during the subject's otherwise planned vitrectomy. The vitrectomy would be started in the usual way, except that the standard modifications would be made for an undiluted vitreous biopsy as discussed above. A 0.2 mL sample would be obtained during the vitreous biopsy. This is the smallest sample the hospital laboratory can analyze and is smaller than what is typically obtained during an undiluted vitreous biopsy.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age, diagnosed to have epiretinal membrane, macular hole, or vitreomacular traction, Otherwise would be needing to undergo vitrectomy procedure

Exclusion Criteria:

* Children & pregnant female Vitrectomy for foreign body extraction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Clinic
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Vitreous Chemistry Analysis | Baseline
  Collection of Vitreous to gain a better understanding of its solute chemistry and the normal relationship of that chemistry to the chemistry of the systemic circulation in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Dara Koozekanani, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States